CLINICAL TRIAL: NCT06368037
Title: To Evaluate the Safety and Feasibility of the DragonFire Transcatheter Radiofrequency Myocardial Ablation System
Brief Title: Feasibility Study of the DragonFire for Hypertrophic Obstructive Cardiomyopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Valgen Medtech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DragonFire-02
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The treament of DragonFire Transcatheter myocardial ablation system (Experimental): If drug therapy does not work or drug side effects are not tolerated, transaortic interventional surgery can be evaluated
  Interventions: Device: DragonFire Transcatheter Myocardial Radiofrequency Ablation System

INTERVENTIONS:
Device: DragonFire Transcatheter Myocardial Radiofrequency Ablation System — The patients with hypertrophic obstructive cardiomyopathy were treated with a transcatheter myocardial radiofrequency ablation system and its guiding system under the guidance of echocardiography

SUMMARY:
This study is a prospective, single-center, single-group design exploratory clinical research. No control group is set, and only subjects meeting the indications of the study device are treated. After patients sign informed consent, they are screened, and those meeting the inclusion criteria are enrolled. The treatment involves using myocardial radiofrequency ablation system and catheter-based myocardial radiofrequency ablation needle and its guidance system for treating obstructive hypertrophic cardiomyopathy. All subjects are followed up before discharge, and at 30 days, 3 months, 6 months, and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥18 years; (2) Diagnosis of obstructive hypertrophic cardiomyopathy, with a peak left ventricular outflow tract gradient (LVOTG) ≥50mmHg at rest or with provocation; (3) Significant clinical symptoms including fatigue, dyspnea, exertional angina, syncope, severely affecting quality of life, and either inadequate response to standardized drug therapy or inability to tolerate drug side effects, with anatomical suitability for alcohol septal ablation and myocardial radiofrequency ablation system and use of catheter-based myocardial radiofrequency ablation needle and its guidance system; (4) NYHA functional class ≥III, or NYHA functional class II patients with one of the following: ① Severe progressive pulmonary arterial hypertension caused by outflow obstruction or resulting mitral regurgitation; ② Atrial fibrillation with associated left atrial enlargement; ③ Exercise treadmill testing indicating reduced cardiac function due to outflow obstruction; (5) Judged by the local clinical trial institution research team as high surgical risk (recommended reference criteria: advanced age or severe comorbidities, or presence of other surgical high-risk factors, such as: ≥2 moderate to severe frailty indicators or potential surgical obstacles, or ≥1 major organ dysfunction that cannot be improved after surgery, or other surgical high-risk factors judged by the cardiac team), or patients who, after being fully informed of the risks and benefits of surgery by the research team, still refuse to undergo surgery; (6) Expected survival of more than 12 months and able to adhere to the follow-up plan; (7) The subject has been informed of the nature of the study, understands the purpose of the clinical trial, voluntarily participates, and signs the informed consent form.

Exclusion Criteria:

* (1) Non-obstructive hypertrophic cardiomyopathy and end-stage hypertrophic cardiomyopathy; (2) Interventricular septum thickness <15mm; (3) Significant diffuse thickening of the interventricular septum; (4) 5-year sudden cardiac death risk score (SCDI) ≥10%, or history of cardiac sudden death (SCD) events, or ventricular fibrillation, or sustained ventricular tachycardia leading to loss of consciousness, or ventricular arrhythmias causing hemodynamic instability in patients without an implanted ICD; (5) Left ventricular ejection fraction <50%; (6) Transthoracic echocardiography suggesting the presence of intracavitary masses, thrombi, or vegetations; (7) History of surgical septal myectomy, alcohol ablation, or other interventricular septal ablation procedures; (8) Any cardiovascular intervention within 30 days or cardiac surgery within 6 months; (9) Concurrent presence of other cardiac diseases requiring surgical treatment, such as severe mitral valve disease, multi-vessel coronary artery disease, etc.; (10) Acute heart failure (defined as acute hemodynamic abnormalities occurring on the basis of primary cardiac or non-cardiac diseases, resulting in a clinical syndrome primarily characterized by acute pulmonary edema, cardiogenic shock, and elevated plasma levels of B-type natriuretic peptide) or end-stage heart failure (defined as resting heart failure, intractable pulmonary edema, or pleural or pericardial effusion despite intensified anti-heart failure treatment); (11) Preoperative presence of right bundle branch block, left bundle branch block, or atrioventricular block requiring permanent pacemaker implantation, or previously implanted permanent cardiac pacemaker; (12) Significant coronary artery disease or critical lesions requiring revascularization due to coronary perfusion-demand mismatch (QFR or FFR <0.8), or those experiencing ischemic events within 30 days; (13) Vascular diseases affecting access for investigational devices, such as aortic aneurysm, severe aortic stenosis, severe aortic arch or aortic valve calcification, or tortuosity or stenosis of the iliac artery; (14) Inability to determine target septal branch or balloon not being fixable in the septal branch, or cardiac anatomy unsuitable for alcohol septal ablation; (15) Hemodynamic instability, defined as systolic blood pressure <90mmHg without the use of afterload-reducing drugs accompanied by symptoms of hypoperfusion, or cardiogenic shock; or requiring vasopressor therapy; or requiring intra-aortic balloon counterpulsation; or other hemodynamic support devices; (16) History of acute peptic ulcer or gastrointestinal bleeding within 3 months; (17) Severe chronic obstructive pulmonary disease (COPD) (requiring continuous home oxygen therapy or long-term use of corticosteroids); (18) History of ischemic cerebrovascular accident (within the past 30 days), or severe carotid artery stenosis (ultrasound showing unilateral carotid artery stenosis >70%), or carotid artery stent implantation within 30 days, or history of hemorrhagic cerebrovascular accident (within 6 months); (19) Bleeding disorders or coagulation disorders, or contraindications to antithrombotic therapy; (20) Renal insufficiency (serum creatinine >2.0mg/dL or 177 µmol/L or eGFR <30 mL/min/1.73m2 or undergoing dialysis treatment; (21) Active infection requiring concurrent antibiotic therapy (if temporary, patients must discontinue antibiotic use for at least 14 days before enrollment); (22) Planned pregnancy, pregnant, or lactating females; (23) Contraindications to transesophageal echocardiography or general anesthesia; (24) Expected lifespan less than 12 months, or disease that would make evaluation of treatment difficult (such as cancer, severe metabolic diseases, psychiatric disorders, etc.) unable to complete the study as required, or poor compliance as judged by the researcher; (25) Currently participating in another experimental drug or medical device clinical study with unfinished primary endpoints or clinical studies that may interfere with the endpoints of this study; (26) Other circumstances judged by the researcher as unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The rate of freedom from major adverse events at 30 days postoperatively | 30 days
  Definition of major adverse events: All-cause mortality within 30 days postoperatively, cardiovascular events requiring emergency intervention, malignant arrhythmias, new indication for permanent pacemaker implantation (non-reversible second-degree type II, high-degree, and third-degree atrioventricular block), left bundle branch block, right bundle branch block.
The success rate of treatment at 6 months postoperatively | 6 months
  Definition of treatment success: Freedom from cardiac death at 6 months postoperatively, freedom from secondary re-intervention due to insufficient reduction in LVOTG, peak left ventricular outflow tract gradient (LVOTG) <30mmHg (at rest) or ≥50% decrease compared to baseline peak LVOTG (at rest or with provocation).

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Phd, Principal Investigator — Northern Theater Command General Hospital of the Chinese People's Liberation Army
Locations (1):
- Northern Theater Command General Hospital of the Chinese People's Liberation Army, Shenyang, China

IPD SHARING:
Plan to Share IPD: No